CLINICAL TRIAL: NCT03963531
Title: Patterns of Care and Outcomes of Patients With METAstatic BONE Tumors in a Real-life Setting
Brief Title: Patterns of Care and Outcomes in Patients With Metastatic Bone Tumors (METABONE)
Acronym: METABONE
Status: Completed | Type: Observational
Sponsor: Institut Bergonié (Other)
Collaborators: French Sarcoma Group (Other)
Responsible Party: Sponsor
Other Study IDs: IB2019-METABONE
Record Dates: First submitted 2019-05-23; First posted 2019-05-24 (Actual); Results first posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Bone Tumor
MeSH Terms: conditions — Bone Neoplasms | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Metastatic Osteosarcoma: Patients aged ≥ 12 years 1/ with a diagnosis of osteosarcoma made by an expert pathologist from one of the French network centers (RESOS), 2/ with an initial diagnosis made from 2008 to 2018, 3/ with a metastatic disease (either synchronous or metachronous), 4/ treated in one of the 11 participating national reference centers designated by the French National Cancer Institute for the management of bone sarcomas
  Interventions: Other: Any cancer treatment
- Metastatic chondrosarcoma: Patients aged ≥12 years (1) with a diagnosis of chondrosarcoma made by an expert pathologist from one of the French network centers, (2) with an initial diagnosis made from 2008 to 2018, (3) with a metastatic disease (either synchronous or metachronous), (4) treated in one of the nine participating national reference centers designated by the French National Cancer Institute for the management of bone sarcomas
  Interventions: Other: Any cancer treatment
- Metastatic Ewing's sarcoma: Patients aged ≥12 years 1/ with a diagnosis of Ewing sarcoma made by an expert pathologist from one of the French network centers (RESOS), 2/ with a diagnosis made from 2008 to 2018, 3/ with a metastatic disease (either synchronous or metachronous ), 4/ treated in one of the 10 national reference centers designated by the French National Cancer Institute for the management of bone sarcomas
  Interventions: Other: Any cancer treatment

INTERVENTIONS:
Other: Any cancer treatment — chemotherapy, surgery, radiotherapy, interventional radiology.
  Other Names: intervention as per recommendations

SUMMARY:
Bone tumors make up about 3-5% of childhood cancers and less than 1% of cancers in adults. Of these, osteosarcoma (OSS) is the most commonly diagnosed primary malignant bone tumor. OSS is a primary mesenchymal malignant tumor of bone characterized by the production of osteoid or immature bone by the malignant cells. Despite its rarity, OSS is the most common primary malignancy of bone in children and adolescents, and the fifth most common malignancy among adolescents and young adults aged 15 to 19 years.

Ewing sarcoma (ES) is the second most frequent bone tumors in children and may arise also in soft tissues. This disease encompasses tumors formerly known as Askin's tumor, Peripheral Neuroectodermal Tumor (PNET) and the Ewing Sarcoma Family of Tumors (ESFT).

Chondrosarcoma are rare sarcoma reputed chemorefractory in the non-operable setting and for which little is known in terms of palliative management with systemic treatments.

Despite adequate loco-regional treatment, up to 40% of patients with sarcoma, soft tissue or bone, will develop metastatic disease. When metastases are detected, the standard of care is based on palliative chemotherapy with a median survival in this setting of only 18 months.

A slight improvement has been obtained over years thank to registration of a couple of drugs such as Trabectedin and Pazopanib, the first antiangiogenic registered for soft tissue sarcoma patients. Pazopanib is routinely prescribed worldwide after failure of first line chemotherapy in soft tissue sarcoma. However, bone tumors have not benefited from these small advances yet and treatment still rely on chemotherapy combining doxorubicine cisplatinum and ifosfamide. There is no standard in relapse and palliative settings, and after failure of these agents the survival is very poor. Bone sarcomas are therefore tumors with very little available data and low level of evidence on palliative systemic treatments in clinical trials and in the real life setting.

The primary objective of the METABONE study is to conduct a retrospective descriptive analysis of clinic-biological profiles, patterns of care and modalities of treatment for a set of patients with malignant bone tumors in a real-life national setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >= 12 years
* Informed consent obtained for inclusion in the databases
* Histology of Ewing's sarcoma type, osteosarcoma, chondrosarcoma
* Diagnostic between 2008 and 2018

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with the diagnosis of Ewing's sarcoma, osteosarcoma, chondrosarcoma,
Sampling Method: Non-Probability Sample
Enrollment: 545 (Actual)
Dates: Start 2008-01-05 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2025-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maud Toulmonde, MD, Principal Investigator — Institut Bergonié
Locations (1):
- Institut Bergonié, Comprehensive Cancer Center, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ducrot C, Dinart D, Reich M, Piffoux M, Bonneau M, Larroquette M, Nannini S, Berchoud J, Bellio H, Cherrier G, Narciso B, Le Cesne A, Bompas E, Gantzer J, Valentin T, Anract P, de Percin S, Boudou-Rouquette P, de Pinieux G, Gouin F, Brahmi M, Bellera C, Toulmonde M. Metastatic chondrosarcoma, patterns of care, and outcomes of patients in a real-life national setting over a decade. Int J Cancer. 2025 Dec 1;157(11):2325-2333. doi: 10.1002/ijc.70023. Epub 2025 Jul 24. PMID 40705468

RESULTS

PARTICIPANT FLOW:
Groups:
- Ewing's Sarcoma: Any cancer treatment: chemotherapy, surgery, radiotherapy, interventional radiology.
Period: Overall Study
Arm/Group | Metastatic Osteosarcoma | Metastatic Chondrosarcoma | Ewing's Sarcoma
Started | 262 | 127 | 156
Completed | 262 | 127 | 156
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metastatic Osteosarcoma | Metastatic Chondrosarcoma | Ewing's Sarcoma | Total
Number analyzed (Participants) | 262 | 127 | 156 | 545
Age, Continuous [Median (Full Range); unit: years] | 27 [12 to 86] | 63 [19 to 90] | 21 [12 to 86] | 40 [12 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 43 | 44 | 199
  Male | 150 | 84 | 112 | 346
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 262 | 127 | 156 | 389

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Interval between the diagnosis of metastatic disease or the first-line systemic therapy onset and the time of death.
Time Frame: 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Metastatic Osteosarcoma | Metastatic Chondrosarcoma | Ewing's Sarcoma
Number analyzed (Participants) | 262 | 127 | 156
months | 21.5 [18.9 to 27.0] | 12.7 [8.2 to 14.9] | 26.6 [21.0 to 32.0]

2. Primary Outcome: Time to Next Treatment (TNT)
Description: time from the systemic treatment onset to the next treatment or death due to any cause, whichever comes first
Time Frame: 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Metastatic Osteosarcoma | Metastatic Chondrosarcoma | Ewing's Sarcoma
Number analyzed (Participants) | 262 | 127 | 156
months | 8.2 [6.7 to 9.9] | 4.6 [3.0 to 5.9] | 12.5 [10.4 to 15.6]

ADVERSE EVENTS:
Time Frame: 5 years Serious and non-serious adverse events were not recorded for the purpose of this study.
Description: Serious and non-serious adverse events were not recorded for the purpose of this study.
Arm/Group | Metastatic Osteosarcoma | Metastatic Chondrosarcoma | Ewing's Sarcoma
All-Cause Mortality (participants affected / at risk) | 172/262 | 93/127 | 115/156
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2007-01-05): https://cdn.clinicaltrials.gov/large-docs/31/NCT03963531/Prot_SAP_000.pdf